CLINICAL TRIAL: NCT01252212
Title: Adherence, Improvement Measure (AIM) System; Challenge Topic: 10-MH-101
Brief Title: Adherence, Improvement Measure (AIM) System
Acronym: AIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The Commonwealth Fund (Other); National Institute of Mental Health (NIMH) (NIH); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-00019; 1RC1MH088341 (NIH)
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Patient Compliance; AIDS
Keywords: HIV, antiretroviral, adherence, SMS, cell phone
MeSH Terms: conditions — Patient Compliance; Acquired Immunodeficiency Syndrome | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receiving SMS alerts (Experimental): The patients randomized to this arm will have a SMS message sent to them regarding medication adherence for antiretroviral medications, anti-hypertensive medications, anti-depressants, hyperglycemic controlling medications and hypercholesterolemia controlling medications as well as life style supportive suggestions.
  Interventions: Behavioral: SMS medication adherence
- No SMS messages (Active Comparator): The patients randomized to this arm will have a SMS message sent to them regarding healthy life style supportive suggestions.
  Interventions: Behavioral: No SMS adherence reminder

INTERVENTIONS:
Behavioral: SMS medication adherence — SMS messages to cell phones.
  Other Names: mobile health messages for health conditions and medications
  Arms: Receiving SMS alerts
Behavioral: No SMS adherence reminder — In this arm, patients will be sent supportive lifestyle suggestions to their phone using SMS technology but will not be sent a reminder regarding their medication adherence.
  Other Names: No medication adherence or disease specific messages.
  Arms: No SMS messages

SUMMARY:
In this project, we will work directly with underserved patients in a safety-net setting to conduct a randomized clinical trial of standard-of-care adherence counseling versus a novel adherence intervention embedded in an existing PHR that uses cellular phone short message service (SMS) reminders and patient responses to the reminders. We will compare adherence rates in both arms as assessed by antiretroviral medication concentrations in hair samples and self-report; clinical outcomes will also be compared in the two arms. The project will examine medication adherence for antiretroviral medications and treatments of common conditions such as depression, hypertension, diabetes and hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18
* Evidence of HIV-1 infection, based on patient's medical history or results of laboratory tests
* Detectable Viral Load, based on patient's medical record
* Receiving primary medical care at the AIDS Program at SFGH
* Able and willing to give informed consent to be randomized to study arms
* Willing to use the patient portal
* Has a cell phone with ability to receive and send unlimited SMS texts, Patient of the HIV/AIDS Clinic at ward 86, SFGH

Exclusion Criteria:

Failure to meet inclusion criteria

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HIV viral load | 12 month
  The primary analyses of the 12-month trial data will compare the two study groups with respect to (i) change from baseline in CD4 T-cell count; and (ii) proportion of patients whose HIV viral load (VL) level is detectable. We will use repeated-measures analysis techniques to estimate longitudinal prevalence at the population level (via generalized estimating equations) and at the individual levels (via generalized linear mixed models)[25].

SECONDARY OUTCOMES:
Level of antiretroviral medication in hair | 12 month
  We will evaluate the antiretroviral level in hair samples from patients to determine compliance with medications.

CONTACTS AND LOCATIONS:
Overall Officials: James Kahn, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Ward 86, San Francisco General Hospital, San Francisco, California, United States